CLINICAL TRIAL: NCT00732433
Title: Digital Mammography: Computer-Aided Breast Cancer Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Heang-Ping Chan Ph.D, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000-0227 HUM 42465
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Tumors, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- digital mammogram (Experimental): Digital mammography is a non-invasive imaging technique to obtain an x-ray image of the breast.
  Two-view digital mammogram of the breast with a lesion that has been recommended for biopsy during the subject's regular clinical care. The digital mammogram is then analyzed by a computer program.
  Interventions: Procedure: digital mammography

INTERVENTIONS:
Procedure: digital mammography — Using non-invasive digital mammography with computer aided programs to screen, detect and characterize breast lesions/cancer.

SUMMARY:
The purpose of this study is to develop computer programs to assist radiologists in finding breast cancer on mammograms and to compare the computer's accuracy of detecting cancers on direct digital and film mammograms.

DETAILED DESCRIPTION:
To develop a computer-aided diagnosis (CAD) system for full field digital mammography (FFDM) using advanced computer vision techniques and to evaluate the effects of CAD on interpretation of digital mammograms (DMs). This system will assist radiologists with the four most important areas in mammographic interpretation: (1) detection of masses, (2) classification of masses, (3) detection of microcalcifications, (4) classification of microcalcifications. The proposed approach is distinctly different from previous approaches in that image information from two-view and bilateral mammograms will be fused with that from the single-view mammogram to improve lesion detection and characterization.

ELIGIBILITY:
Inclusion Criteria:

* Females who have been scheduled for mammographic exams.
* Females who have been recommended for work-up or biopsy due to a suspicious finding on their mammogram.
* Females who can give informed consent.

Exclusion Criteria:

* No subject under 18 years of age

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2000-06 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Using computer aided programs to assist in detection and characterization of breast lesions in digital mammography. | Research scan will be completed at the time of scheduled clinical visit.

CONTACTS AND LOCATIONS:
Overall Officials: Heang-Ping Chan, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States